CLINICAL TRIAL: NCT06590337
Title: Radicle Spark for Men™ 24: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Sexual Health and Related Health Outcomes
Brief Title: Radicle Spark for Men 24: A Study of Health and Wellness Products on Sexual Health and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2413
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-11

CONDITIONS: Sexual Satisfaction; Sexual Function
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their age and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' study product assignment. Participants are blinded to the study product they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control 1 (Placebo Comparator): Spark Product Form 1 - control
  Interventions: Dietary Supplement: Spark Placebo Control Form 1
- Active Product 1.1 (Experimental): Spark Product Form 1 - active product 1
  Interventions: Dietary Supplement: Spark Active Study Product 1.1 Usage
- Placebo Control 2 (Placebo Comparator): Spark Product Form 2 - control
  Interventions: Dietary Supplement: Spark Placebo Control Form 2
- Active Product 2.1 (Experimental): Spark Product Form 2 - active product 1
  Interventions: Dietary Supplement: Spark Active Study Product 2.1 Usage

INTERVENTIONS:
Dietary Supplement: Spark Placebo Control Form 1 — Participants will use their Radicle Spark Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Spark Active Study Product 1.1 Usage — Participants will use their Radicle Spark Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Spark Placebo Control Form 2 — Participants will use their Radicle Spark Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Spark Active Study Product 2.1 Usage — Participants will use their Radicle Spark Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1

SUMMARY:
A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on sexual health and related health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants. residing in the United States.

Eligible participants will (1) endorse a desire for improved libido, sexual satisfaction and/or function, (2) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities: Assigned sex at birth is male
* Resides in the United States
* Endorses as improved libido (sex drive), sexual satisfaction and/or function as a primary desire
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients: NYHA (New York Heart Health) Class Ill or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy. immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOls (monoamine oxidase inhibitors), or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned sex at birth is male
Enrollment: 1202 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in sexual health | 6 weeks
  Difference between rates of change over time in sexual health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Brief Profile Sexual Function and Satisfaction Survey [male version consists of 4 health domains assessed only among participants with sexual activity in the 30 days prior: erectile function (score range = 2-10; higher scores indicate better erectile function), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]

SECONDARY OUTCOMES:
Change in feelings of stress | 6 weeks
  Mean difference in feelings of stress score as assessed by Perceived Stress Scale 4 (PSS-4) (scale 0-16; where lower scores correspond to less stress)
Change in fatigue | 6 weeks
  Mean difference in fatigue as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in mood score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; where higher scores correspond to more severe emotional distress-depression)
Minimal clinical importance difference (MCID) in sexual health | 6 weeks
  Likelihood of achieving a MCID in sexual health score as assessed by Patient Reported Outcome Measurement System (PROMIS) Brief Profile Sexual Function and Satisfaction Survey [male version consists of 4 health domains assessed only among participants with sexual activity in the 30 days prior: erectile function (score range = 2-10; higher scores indicate better erectile function), orgasm ability (score range = 1-5; higher scores indicate more ability), orgasm pleasure (score range = 1-5; higher scores indicate more pleasure), satisfaction with sex life (score range = 2-10; higher scores indicate more satisfaction)]
Minimal clinical importance difference (MCID) in feelings of stress | 6 weeks
  Likelihood of achieving a MCID in feelings of stress score as assessed by Perceived Stress Scale 4 (PSS-4) (scale 0-16; where lower scores correspond to less stress)
Minimal clinical importance difference (MCID) in fatigue | 6 weeks
  Likelihood of achieving a MCID in feelings of fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Minimal clinical importance difference (MCID) in mood (emotional distress-depression) | 6 weeks
  Likelihood of achieving a MCID in mood score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; where higher scores correspond to more severe emotional distress-depression)

OTHER OUTCOMES:
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (1) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based IgG (Immunoglobulin) biomarker (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (2) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based cytokines (Interleukin 1 beta, Interleukin 8, Tumor necrosis factor-alpha, and Interleukin 6) biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (3) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based dehydroepiandrosterone sulfate (DHEA-S) biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (4) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based estradiol biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (5) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based progesterone biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (6) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based testosterone biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (7) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based cortisol biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (8) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based melatonin biomarker. (Optional; among consented participants only).
Change in saliva concentration of at-home (direct-to-consumer) specimen assay (9) | 6 weeks
  Mean difference in saliva concentration as assessed by saliva-based C-Reactive Protein (CRP) biomarker. (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (1) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based cortisol biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (2) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based homocysteine biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (3) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based ferritin biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (4) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based thyroid stimulating hormone (TSH) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (5) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based hemoglobin A1C (HbA1c) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (6) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based insulin biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (7) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based vitamin D biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (8) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based dehydroepiandrosterone sulfate (DHEA-S) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (9) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based testosterone biomarker (1 drop) (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (10) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based estradiol biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (11) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based total cholesterol (high-density lipoproteins (HDL) and low-density lipoproteins (LDL)) biomarker (1 drop). (Optional; among consented participants only).
Change in blood concentration of at-home (direct-to-consumer) specimen assay (12) | 6 weeks
  Mean difference in blood concentration as assessed by blood-based triglycerides (apolipoprotein A1 (ApoA1) and apolipoprotein B (ApoB)) (1 drop). (Optional; among consented participants only).
Change in stool concentration of at-home (direct-to-consumer) specimen assay | 6 weeks
  Mean difference in stool concentration as assessed by a stool sample (microbial diversity) (Optional; among consented participants only).

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com